CLINICAL TRIAL: NCT02694614
Title: Weight-loss Treatment of Overweight / Obesity Patients Through Smartphone-assisted Dietary Coaching: A Pre-post Pilot Study
Brief Title: Weight-loss Treatment Through Smartphone-assisted Dietary Coaching
Acronym: Oviva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oviva AG (Industry)
Collaborators: Bern University of Applied Sciences (Other); Zentrum für Adipositas- und Stoffwechselmedizin Winterthur GmbH (Industry); Swiss Commission for Technology and Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17236.2 PFLS-LS
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Overweight; Obesity
Keywords: weight loss; individualised dietary coaching; smartphone-assisted dietary coaching; health behavior change
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- smartphone-assisted dietary coaching (Experimental)
  Interventions: Behavioral: smartphone-assisted dietary coaching

INTERVENTIONS:
Behavioral: smartphone-assisted dietary coaching

SUMMARY:
The purpose of this study is to evaluate the effectiveness and feasibility of weight loss counselling via a smartphone-app for patients with overweight/obesity in a 1-year long pilot study.

The study is organized in the following phases:

Recruitment (-14 to -2). Participants will be informed about the study. Participants agreed to enter the study and signed an informed consent.

Screening / Baseline measurement (week -2) Inclusion criteria will be checked. Anthropometric measurements: height, weight, waist circumference, body fat, blood pressure measurement, blood sampling for blood glucose; HbA1c, Insulin; Triglyceride, HDL-Cholesterol (assessment Part I). During the visit participants are requested to fill in a paper-pencil questionnaire: socioeconomic background (only at the beginning of the study), dietary and exercise habits, health-related quality of life, self-effectiveness (assessment part II). The participants are introduced to the smartphone assisted coaching.

Introductory phase (2 weeks): Participants take pictures of their meals with the app, which they send to the dietitian. After the introductory phase, the patients and the dietitians discuss via app how the patients should change their habits and agree on goals to reduce their weight.

Phase 1 (12 weeks): Intensive online counselling with the smartphone app, with the agreed upon goals in mind (5 days per week + one Skype call). Group counselling session with / without a dietitian are held if necessary. Furthermore, the dietitians make available information material for patient specific dietary topics online. Week 12: assessment I+II.

Phase 2 (until week 25): The habits that further a weight reduction are being stabilised - the frequency of the online counselling is reduced (3 days per week), group counselling with / without a dietitian are held if necessary. Furthermore, the dietitians hand out information material for patient specific dietary topics.

Phase 3 (week 26-52): This phase is relevant for maintaining the patient's wright. Online counselling happens once every 2 weeks. Group counselling with / without a dietitian are held if necessary. Furthermore, the dietitians hand out information material for patient specific dietary topics. At the end end, the dietitians will again collect data (assessment I+II). The online counselling process is evaluated with 3 group discussions.

Follow-up (week 104)

DETAILED DESCRIPTION:
Recruitment process will be conducted in two parts. During the first part potential participants will be recruited:

* At the obesity centre during the current obesity consultation
* During regularly information events at the obesity centre flyers will be handed out.
* During training courses for general practitioner at the obesity centre flyers will be handed out.
* Through the network Medical AdiNetwork flyers will be send to general practitioner.
* Advertisement: via website Oviva, Berne University of Applied Science, Zentrum für Adipositas- und Stoffwechselmedizin Winterthur (ZAS) GmbH; Newspaper "Winterthur Stadt Anzeiger".

Participants receive written and verbal information about the study. After participants have given informed consent for participation the second phase (screening process) take place. The researchers determine eligibility of participants based on the inclusion and exclusion criteria at the Zentrum für Adipositas- und Stoffwechselmedizin Winterthur GmbH.

Description of variables:

Weight: Measurement take place in the morning, using a clinically validated and calibrated scale (Seca mBCA 515, medical Body Composition Analyzer). The participant should be clothed lightly, without shoes. Weight is recorded within 0.01 kg.

BMI is calculated by dividing body weight (in kilograms) by height (in meters)2 Height is measured using a calibrated stadiometer (Forma Seca). The subject stands erect with feet positioned on the floor board of the stadiometer. Heels, buttocks, and back of head touch the back board of the stadiometer with arms by sides.

Waist circumference: For the measurement the tape will be located midway between the lower rib and iliac crest. Each measurement is performed twice and recorded within 0.5 cm. If the difference between the measurements is greater than 1 cm, a third measurement will be performed, and the mean of the two closest measurements will be calculated. The participant stand with feet close together, wear little clothing, should be relaxed, and the measurements should be taken at the end of a normal expiration.

Body fat will be measured by Bioelectrical impedance analysis (Seca mBCA 515, medical Body Composition Analyzer). Participants will be asked not to eat, not to drink, not to smoke and not to do any sport 1h before BIA measurement. They were also asked not to consume caffeine or alcohol and other drugs 24 hours before. Bladder should be emptied before measurement. Participants are lightly dressed during measurement and wear no tights. Measurement while Standing.

Laboratory parameters: Subjects have to be fasting over night (8 hours), abstained from smoking, alcohol ingestion, caffeine-containing beverages, and vigorous exercise 48 h before the experiments. The investigators inserted one venous catheter in a large antecubital vein for blood sampling at week 0, 12 and 52.

Blood glucose: filling in a small fluoride containing tube to put aside in the refrigerator at 5°C. Standard value: < 5.6 mmol/l.

HbA1c: filling in a small EDTA containing tube to put aside in the refrigerator at 5°C. Standard value: <5.6%.

Triglyceride: filling in a special tube for centrifugation (10 min at 6000 rpm) for extraction of blood serum to put aside in the refrigerator at 5°C. Standard value: < 2.26 mmol/l.

Insulin: filling in a special tube for centrifugation (10 min at 6000 rpm) for extraction of blood serum to put aside in the refrigerator at 5°C. Standard value: 2.6-24.9 mIU/l.

HDL-Cholesterol: filling in a special tube for centrifugation (10 min at 6000 rpm) for extraction of blood serum to put aside in the refrigerator at 5°C. Standard value: > 1.69 mmol/l (no cardiovascular risk); 1.15-1.68 mmol/l (moderate cardiovascular risk); < 1.14 mmol/l (high cardiovascular risk)

Beta-HCG filling in serum tube with seperating gel. Standard value: <5 U/I.

Vital signs: Blood pressure and heart rate will be investigated by the method of Riva Rocci with a special measuring instrument (Firma boso-medicus SN 768 00 440 729 Bosch+Sohn GmbH und Co) and a stethoscope. The patient has to be sit down for more then 15 min. These measurements will be carried out 3 times in a row and the mean value will be used.

Statistical Analysis

The following statistical hypotheses will be tested for the primary outcome:

Null hypothesis: Change in weight from baseline to week 52 = 0 Alternative hypothesis: Change in weight from baseline to week 52 ≠ 0 The sample size calculation was based on the statistical hypotheses. Using a two-sided Wilcoxon signed-rank test with significance level 0.05 and power 80%, a sample size of 36 is needed to detect a weight change from baseline to week 52 of 0.5 standard deviation, which corresponds to a medium effect size according to Cohen. To account for drop-outs 50 patients will be enrolled in the study

The following analysis populations will be used:

* Intention-to-treat (ITT) Population.
* Per protocol (PP) Population.

The primary outcome will be analyzed based on the ITT population. A supportive analysis based on the PP population will be performed. For the primary outcome, the change in weight will be calculated from baseline to week 52. The null hypothesis will be tested using a two-sided Wilcoxon signed-rank test with significance level 0.05. All outcomes will be analyzed based on the ITT population. Supportive analyses based on the PP population will be performed. For all secondary outcomes the changes will be calculated from baseline to the specified time points. The changes over the whole observation period will be investigated using non-parametric ANOVA methods for longitudinal data. Post-hoc tests for changes at all measured time points may be performed using Wilcoxon signed-rank tests. Correlations between outcome variables will be investigated using Spearman's rank correlation coefficient. Two-tailed tests with significance level 0.05 will be used for all analyses. No adjustment for multiple testing will be performed. All outcome variables will be summarized using descriptive statistics. All analyses will be performed using the latest version of R (http://www.r-project.org).

No imputation of missing data will be performed. A row denoted "Missing" will be included in count tabulations if necessary to account for drop-outs and missing values. For continuous variables a column with the number of available observations will be added. Patients lost to follow-up before reaching the primary outcome will not be replaced. The expected drop-out rate has been accounted for in the sample size calculation.

Data Management

* for smartphone assisted coaching: Data entry by users (both the patient and the dietitian) are always validated used predefined patterns and range checks. If for any reason something goes wrong the user is informed about the unsuccessful data entry and might be (depending on the severity of the error) forced to login to the respective system again to assert that no inconsistent state is displayed to the user. Data is kept consistent by validity checks defined by dietitians and is stored in a highly structured and consistency-constrained database hosted by a medical infrastructure provider.
* On-site clinical data management: All data are acquired by 2 persons (study nurse and clinical subinvestigator) and are electronically immigrated from different equipment in our electronically database. Data can than extracted for CRF and data analysis. The patient key list will be archived at the clinic site, only the PI has the insight.
* All electronic data will be transferred via secure connections and stored in a secure facility, according to regulations for sensitive private information.

Adverse or serious adverse events are not expected in this kind of intervention. But if happen, these events will be described in the CRF, because they may be happened non-causal.

Quality assurance: All study personnel will be instructed by the PI for all study procedures. The PI will furthermore ensure on-going correct data collection at the obesity center and the Sponsor will ensure Oviva technical functionality and coaching operations. All study data will be archived for a minimum of 10 years after study termination or premature termination of the clinical trial.

Follow standardized procedures and in accordance with the provisions blood samples are generally stored at 5 degree celsius. Default storage: Blood samples (EDTA) for seven days; Blood serum for one year. Afterwards, blood samples are destroyed.

If the subject withdraws consent, the blood samples will be analyzed and afterwards destroyed immediately. Data will be analyzed and anonymised.

Monitoring: The monitor will visit the PI and study centre at periodic intervals, in addition to maintaining necessary telephonic and written communication. The monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the PI and their study team.

* An initiation visit will be performed before starting recruitment to ensure that the site personnel have been thoroughly trained and the site is provided with all clinical trial supplies.
* The first monitoring visit will be conducted in March 2016 shortly after the first participant has been enrolled to ensure that criteria for inclusion and exclusion have been met and that all protocol procedures are being followed appropriately. All patients enrolled will be verified to have met all inclusion criteria.
* Subsequent monitoring visits: Study Site will be monitored approximately 3 times depending on the demands of the study (week 12, week 52, and week 104).
* Closure of Study: A Site Close-Out Visit will be conducted after all participants have completed the study and all queries have been answered. At this visit the monitors will ensure that all trial documentation is in place, and will discuss archiving procedures with the site.
* Communication between visits: Between monitoring visits, investigators will be telephoned regularly by the monitors to verify patient enrolment status, review study progress, answer protocol questions, CRF completion status and queries, and to ensure that the study proceeds in a timely manner.

Change Management: Basically, study will be conducted in compliance with the study protocol. If deviations are necessary, like changes to eligibility criteria, study design, recruitment, assessment, intervention, outcomes, analyses) the proposed amendment will be submitted well-founded to the sponsor. All investigators can make written suggestions in this regard after consulting principal investigator. A written consent will be obtained from the sponsor.

Substantial amendments are only implemented after approval of the CEC. Under emergency circumstances, deviations from the protocol to protect the rights, safety and well-being of human subjects may proceed without prior approval of the sponsor and the CEC. Such deviations will be documented and reported to the sponsor and the CEC as soon as possible.

All Non-substantial amendments are communicated to the CEC within the Annual Safety Report (ASR). Changes in the protocol are performed by the PI. The written correspondence is kept in the Investigator Site File.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Adults (18 years and over; BMI ≥ 27 kg/m2 and ≤ 32 kg/m2) with fluent German
* Smartphone user (iOS or Android)
* Capable of sending / receiving text messages and pictures

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Persons who were on a diet during the last 6 months; take medication for weight loss at any time before, or are enrolled in another weight loss program
* Persons with nutrition therapy dependent diseases and other serious diseases requiring continuous drug therapy
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Individuals who will perform the interventions: registered dietitians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Body weight change | from baseline to week 52

SECONDARY OUTCOMES:
Body weight change | from baseline to week 12, week 104 (follow-up)
BMI Change | from baseline to week 12, week 52, week 104 (follow-up)
Body fat | from baseline to week 12, week 52, week 104 (follow-up)
Waist circumference | from baseline to week 12, week 52, week 104 (follow-up)
HBA1c | from baseline to week 12, week 52, week 104 (follow-up)
Fasting glucose | from baseline to week 12, week 52, week 104 (follow-up)
Fasting insulin | from baseline to week 12, week 52, week 104 (follow-up)
Triglyceride | from baseline to week 12, week 52, week 104 (follow-up)
HDL-cholesterol | from baseline to week 12, week 52, week 104 (follow-up)
Blood pressure | from baseline to week 12, week 52, week 104 (follow-up)
Physical Activity assessed using the Global physical activity Questionnaire (GPAQ) | from baseline to week 12, week 52, week 104 (follow-up)
  To assess changes in physical activity, the investigators will use the Global physical activity Questionnaire (GPAQ)
Eating behaviour assessed using a brief dietary assessment | from baseline to week 12, week 52, week 104 (follow-up)
  To assess changes in eating behavior, the investigators will use a brief dietary assessment
Overall health status assessed using the short version quality of life assessment tool (SF12) | from baseline to week 12, week 52, week 104 (follow-up)
  To assess changes of the overall health status, the investigators will use the short version quality of life assessment tool (SF12)
Self-efficacy assessed using a questionnaire | from baseline to week 12, week 52, week 104 (follow-up)
  To assess the self-efficacy related to dietary change, the investigators will use a questionnaire from Hahn, Schwarzer, Renner (1996)

OTHER OUTCOMES:
Contact frequency with dietician | from baseline to week 12, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Karin Haas, Dr.rer.nat., Study Chair — Bern University of Applied Sciences; Susanne Maurer-Wiesner, Dr.med., Principal Investigator — Zentrum für Adipositas- und Stoffwechselmedizin Winterthur GmbH; Kai Eberhardt, Dr.sci.ETH, Study Director — Oviva AG
Locations (1):
- Zentrum für Adipositas und Stoffwechselmedizin Winterthur GmbH, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Donaldson EL, Fallows S, Morris M. A text message based weight management intervention for overweight adults. J Hum Nutr Diet. 2014 Apr;27 Suppl 2:90-7. doi: 10.1111/jhn.12096. Epub 2013 Jun 6. PMID 23738786
- [Result] Aguilar-Martinez A, Sole-Sedeno JM, Mancebo-Moreno G, Medina FX, Carreras-Collado R, Saigi-Rubio F. Use of mobile phones as a tool for weight loss: a systematic review. J Telemed Telecare. 2014 Sep;20(6):339-49. doi: 10.1177/1357633X14537777. Epub 2014 May 29. PMID 24875928
- [Result] Appel LJ, Clark JM, Yeh HC, Wang NY, Coughlin JW, Daumit G, Miller ER 3rd, Dalcin A, Jerome GJ, Geller S, Noronha G, Pozefsky T, Charleston J, Reynolds JB, Durkin N, Rubin RR, Louis TA, Brancati FL. Comparative effectiveness of weight-loss interventions in clinical practice. N Engl J Med. 2011 Nov 24;365(21):1959-68. doi: 10.1056/NEJMoa1108660. Epub 2011 Nov 15. PMID 22085317
- [Result] Fukuoka Y, Kamitani E, Bonnet K, Lindgren T. Real-time social support through a mobile virtual community to improve healthy behavior in overweight and sedentary adults: a focus group analysis. J Med Internet Res. 2011 Jul 14;13(3):e49. doi: 10.2196/jmir.1770. PMID 21752785
- [Result] Hutchesson MJ, Rollo ME, Krukowski R, Ells L, Harvey J, Morgan PJ, Callister R, Plotnikoff R, Collins CE. eHealth interventions for the prevention and treatment of overweight and obesity in adults: a systematic review with meta-analysis. Obes Rev. 2015 May;16(5):376-92. doi: 10.1111/obr.12268. Epub 2015 Mar 5. PMID 25753009
- [Result] Levine DM, Savarimuthu S, Squires A, Nicholson J, Jay M. Technology-assisted weight loss interventions in primary care: a systematic review. J Gen Intern Med. 2015 Jan;30(1):107-17. doi: 10.1007/s11606-014-2987-6. Epub 2014 Aug 19. PMID 25134692
- [Result] Okorodudu DE, Bosworth HB, Corsino L. Innovative interventions to promote behavioral change in overweight or obese individuals: A review of the literature. Ann Med. 2015 May;47(3):179-85. doi: 10.3109/07853890.2014.931102. Epub 2014 Jul 10. PMID 25011006
- [Result] Radcliff TA, Bobroff LB, Lutes LD, Durning PE, Daniels MJ, Limacher MC, Janicke DM, Martin AD, Perri MG. Comparing Costs of Telephone vs Face-to-Face Extended-Care Programs for the Management of Obesity in Rural Settings. J Acad Nutr Diet. 2012 Sep;112(9):1363-1373. doi: 10.1016/j.jand.2012.05.002. Epub 2012 Jul 19. PMID 22818246
- [Result] Vodopivec-Jamsek V, de Jongh T, Gurol-Urganci I, Atun R, Car J. Mobile phone messaging for preventive health care. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007457. doi: 10.1002/14651858.CD007457.pub2. PMID 23235643
- [Result] Siopis G, Chey T, Allman-Farinelli M. A systematic review and meta-analysis of interventions for weight management using text messaging. J Hum Nutr Diet. 2015 Feb;28 Suppl 2:1-15. doi: 10.1111/jhn.12207. Epub 2014 Jan 31. PMID 24480032
- [Result] Wing RR, Tate DF, Gorin AA, Raynor HA, Fava JL. A self-regulation program for maintenance of weight loss. N Engl J Med. 2006 Oct 12;355(15):1563-71. doi: 10.1056/NEJMoa061883. PMID 17035649
- [Derived] Haas K, Hayoz S, Maurer-Wiesner S. Effectiveness and Feasibility of a Remote Lifestyle Intervention by Dietitians for Overweight and Obese Adults: Pilot Study. JMIR Mhealth Uhealth. 2019 Apr 11;7(4):e12289. doi: 10.2196/12289. PMID 30973338